CLINICAL TRIAL: NCT00868426
Title: Pharmacokinetic Pilot Study on Budesonide/Formoterol Device-metered Dry Powder Inhaler, Symbicort Turbuhaler; an Open, Single Center, Single Dose Study With 3-way Crossover Design in Healthy Subjects
Brief Title: Pharmacokinetic Pilot Study on Budesonide/Formoterol Device-metered Dry Powder Inhaler
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Ulla Sairanen, Clinical study director, Orion Corporation, Orion Pharma
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3103001
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: Healthy volunteer study
MeSH Terms: interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination; Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Budesonide/Formoterol Batch 1
  Interventions: Drug: Budesonide/Formoterol Batch 1
- 2 (Experimental): Budesonide/Formoterol Batch 2
  Interventions: Drug: Budesonide/Formoterol Batch 2
- 3 (Experimental): Budesonide/Formoterol Batch 1 and charcoal
  Interventions: Drug: Budesonide/Formoterol Batch 1 and charcoal

INTERVENTIONS:
Drug: Budesonide/Formoterol Batch 1 — Single, inhaled dose
  Other Names: Symbicort Turbuhaler
  Arms: 1
Drug: Budesonide/Formoterol Batch 2 — Single, inhaled dose
  Other Names: Symbicort Turbuhaler
  Arms: 2
Drug: Budesonide/Formoterol Batch 1 and charcoal — Single, inhaled dose
  Other Names: Symbicort Turbuhaler
  Arms: 3

SUMMARY:
The aim of this pilot study is to assess the methodology, practical arrangements and pulmonary absorption with charcoal blockage for the future bioequivalence studies. In addition, PK of budesonide and formoterol after administration from 2 different batches of Symbicort TH is compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* Good general health ascertained by detailed medical history, and laboratory and physical examinations
* Finnish speaking males and females, 18-55 (inclusive) years of age
* Normal weight defined as body mass index (BMI) > 19 and < 30 kg/m2
* Weight at least 50 kg
* Regular intestinal transit

Exclusion Criteria:

* Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological or psychiatric disease
* Any abnormal value of laboratory, vital signs, 12-lead electrocardiogram or physical exam which may in the opinion of the investigator interfere with the test results or cause a health risk for the subject if he/she takes part into the study
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study
* Known hypersensitivity to the active substance(s) or to any of the excipients of the drug
* Pregnant or lactating females
* Recent or current (suspected) drug abuse or positive result in the drugs abuse test
* Recent or current alcohol abuse (regular drinking more than 21 units per week for males and more than 16 units per week for females [1 unit = 4 cl spirits or equivalent])
* Current use of nicotine containing products more than 5 cigarettes (or equivalent)/day and/or inability to refrain from the use of nicotine containing products during the study
* Use of caffeine containing beverages more than 600 mg of caffeine/day and/or inability to refrain from the use of caffeine containing beverages during the treatment periods until 24 h after study treatment administration
* Blood donation or loss of significant amount of blood within 90 days prior to the first study treatment administration
* Administration of another investigational drug within 90 days prior to the first study treatment administration
* Unsuitable veins for repeated venipuncture or for cannulation
* Inability to learn the correct inhalation technique
* Inability to participate in all treatment periods

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Assess the methodology, practical arrangements and pulmonary absorption with charcoal blockage | 1 day

SECONDARY OUTCOMES:
Pharmacokinetics of budesonide and formoterol after administration of two different batches of Symbicort Turbuhaler | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo Ingman, MD, PhD, Principal Investigator — Orion Corporation, Orion Pharma
Locations (1):
- Orion Pharma Phase I Unit, Espoo, Finland